CLINICAL TRIAL: NCT06732947
Title: AI Integration in Academic Writing: a Study on Qualitative Research in Physical Therapy Education
Brief Title: AI Integration in Academic Writing
Status: Not yet recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, Lecturer, Kafrelsheikh University
Other Study IDs: KFSIRB200-434
Record Dates: First submitted 2024-11-29; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Artificial Intelligence (AI); Qualitative Research
Keywords: AI integrating; academic writing; artificial intellegance; AI in education; AI tools; physical therapy students

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- university students between age of 20 and 22

SUMMARY:
This study aims to explore the effect of AI use on different aspects of writing qualitative research papers by physical therapy students. By examining how AI tools influence various elements of the writing process, such as structure, clarity, knowledge presentation, and critical thinking, this research aims to provide insights into the benefits and potential drawbacks of AI integration in academic assignments. By recognizing the significance of this research, contribute to understanding how AI can be effectively utilized to enhance the educational experience and improve the writing skills of physical therapy students.

DETAILED DESCRIPTION:
This study aims to explore the effect of AI use on different aspects of writing qualitative research papers by physical therapy students. By examining how AI tools influence various elements of the writing process, such as structure, clarity, knowledge presentation, and critical thinking, this research aims to provide insights into the benefits and potential drawbacks of AI integration in academic assignments. By recognizing the significance of this research, contribute to understanding how AI can be effectively utilized to enhance the educational experience and improve the writing skills of physical therapy students.

This study explores how AI can enhance academic writing and analysis in physical therapy education, focusing on how AI tools may support researchers in qualitative work.

This project is significant as it addresses several key benefits and challenges of AI integration in academic writing for qualitative research within physical therapy education:

1. Enhancing academic writing skills and motivation: Quantitative analysis reveals significant improvements in both writing skills and motivation among students who received AI-assisted instruction compared to the control group. The experimental group demonstrates enhanced proficiency in various aspects of writing, including organization, coherence, grammar, and vocabulary.
2. The importance of transparency:The study provides an understanding of the current landscape of declaring the use of generative AI tools by authors in nursing journals. Future studies could examine the implications of such disclosure on reader perception and the evaluation of research quality. This would help shed light on the effectiveness of disclosure in enhancing transparency and trust in academic writing. Furthermore, developing guidelines or best practices for the appropriate declaration of generative AI usage by authors and reviewers would be beneficial in ensuring consistent and responsible implementation of AI technologies in scholarly research.
3. Promising Perspectives and Valid Concerns: The imminent dominant use of LLM technology including the widespread use of ChatGPT in health care education, research, and practice is inevitable. Considering the valid concerns raised regarding its potential misuse, appropriate guidelines and regulations are urgently needed with the engagement of all stakeholders involved to ensure the safe and responsible use of ChatGPT powers. The proactive embrace of LLM technologies with careful consideration of the possible ethical and legal issues can limit the potential future complications.
4. ethical consideration: concerns exist about plagiarism and ghostwriting, the unreliability of results, copyright issues, educational gaps due to technological advancement, and decreased learning ability. Educators are concerned about students' reliance on AI. Using ChatGPT to solve writing or computer coding assignments may hinder students' learning, and New York City public schools have blocked access to ChatGPT on campus.

ELIGIBILITY:
Inclusion Criteria:

* university students between the ages of 20 and 22.

Exclusion Criteria:

* no exclusion criteria

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: kafrelsheikh university students
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
percentage of AI-generated content within the text of each assignment. | During the procedure
Incidence of Structure & Organization (SO) by Sapling AI detector website | During the procedure
  This criterion evaluates the overall layout and logical flow of the research paper. It includes the clarity of the introduction, body, and conclusion, as well as the coherence of arguments and the seamless transition between sections. A well-structured paper should have a clear beginning, middle, and end, with each part contributing to the overall argument or narrative.
Rate Writing Clarity (WC) by Sapling AI detector website | During the procedure
  Writing Clarity assesses the ease with which the reader can understand the text. This includes the use of clear and precise language, the absence of grammatical and typographical errors, and the appropriateness of sentence structure and word choice. A paper with high writing clarity will be easily comprehensible and free from ambiguity
Rate of Knowledge (Know) by Sapling AI detector website | During the procedure
  This criterion measures the depth and breadth of the student's understanding of the subject matter. It includes the accurate representation of key concepts, theories, and research findings related to the topic. A high score indicates that the student has demonstrated a thorough and nuanced understanding of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Reda Fathi Elbosaty, bachelor student, Principal Investigator — Faculty of physical therapy, kafrelsheikh university; Noran Abdallah Essa, bachelor student, Principal Investigator — Faculty of physical therapy, kafrelsheikh university; Ahmed Ali Torad, PhD, lecturer, Principal Investigator — Faculty of physical therapy Kafrelsheikh university; Tamer Mohamed El-Saeed, PhD, associate professor, Study Director — Cairo University
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request from the principal investigator.